CLINICAL TRIAL: NCT03366532
Title: Dietary Analyses in the Nurses' Health Studies and Health Professionals Follow-Up Study (Diabetes, Cardiovascular Disease, and Mortality)
Brief Title: Dietary Analyses in the Nurses' Health Study, Nurses' Health Study II, and Health Professionals Follow-Up Study
Acronym: Diet
Status: Completed | Type: Observational
Sponsor: Harvard School of Public Health (HSPH) (Other)
Collaborators: Harvard Medical School (HMS and HSDM) (Other)
Responsible Party: Principal Investigator, Qi Sun, Associate Professor of Medicine, Harvard School of Public Health (HSPH)
Other Study IDs: 2000-P-002221
Record Dates: First submitted 2017-12-04; First posted 2017-12-08 (Actual); Last update posted 2017-12-08 (Actual); Status verified 2017-12

CONDITIONS: Type2 Diabetes; Coronary Artery Disease; Morality; Stroke
Keywords: diet; food frequency questionnaire; nutrient
MeSH Terms: conditions — Coronary Artery Disease; Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Nurses' Health Study: The NHS began in 1976 when 121,700 female nurses aged 33-55 years and residing in the United States responded to a baseline questionnaire.
  Interventions: Other: Dietary assessments
- Nurses' Health Study II: The NHSII was initiated in 1989 with the recruitment of 116,671 younger female registered nurses, 24 to 44 years of age, from 14 states
  Interventions: Other: Dietary assessments
- Health Professionals Follow-Up Study: The Health Professionals Follow-up Study (HPFS) was established in 1986 and was comprised of 51,529 US male health professionals ranging in age from 40 to 75 years at enrollment from 50 states
  Interventions: Other: Dietary assessments

INTERVENTIONS:
Other: Dietary assessments — We use food frequency questionnaires to collect and update intake of foods and nutrients in observational studies. No intervention is involved.

SUMMARY:
To determine the relationships of a variety of nutrients, foods, and dietary patterns with the subsequent risk of developing type 2 diabetes, cardiovascular disease, and mortality in US men and women.

DETAILED DESCRIPTION:
The Nurses' Health Study (NHS) consisted of 121,700 female registered nurses aged 30 to 55 years from 11 US states who were enrolled in 1976. The NHSII was initiated in 1989 with the recruitment of 116,671 younger female registered nurses, 24 to 44 years of age, from 14 states. The Health Professionals Follow-up Study (HPFS) was established in 1986 and was comprised of 51,529 US male health professionals ranging in age from 40 to 75 years at enrollment from 50 states.

Study investigators sent follow-up questionnaires biennially to participants to update information on past medical history as well as lifestyle factors. Validated food frequency questionnaires (FFQs) were first sent in 1980 for the NHS, 1991 for the NHSII, and 1986 for the HPFS. Dietary assessments have been updated every 2-4 years since baseline. The FFQs collect information on average intake of each food item over the past year. It also specifies a common serving size for each item. Participants could select from one of nine intake frequency choices, ranging from less than once per month to six or more times per day. Participants also provided information on current use and dose of multivitamins and use of other vitamin supplements.

For these three cohorts, investigators repeatedly collected and updated information on several anthropometric and lifestyle factors such as weight, smoking status, alcohol use, coffee intake, and physical activity level. Information was also collected on several major risk factors.

Study subjects reported new diagnoses biennially. After obtaining permission from participants, their medical and pathological records were acquired. Study physicians blinded to questionnaire information reviewed these records to confirm diagnoses of coronary heart disease and stroke. Self-reported diabetes diagnoses are confirmed using a validated supplementary questionnaire on symptoms, blood glucose levels, and medication use. Deaths are identified through reports from next of kin, postal authorities, or by searching the National Death Index.

All investigations regarding dietary factors in relation to type 2 diabetes, cardiovascular disease, and mortality have been approved by the institutional review boards of both Brigham and Women's Hospital and Harvard T.H Chan School of Public Health.

ELIGIBILITY:
Inclusion Criteria:

* Returned baseline food frequency questionnaires (FFQs).

Exclusion Criteria:

* Participants who had died or reported a diagnosis of diabetes (including type 1 diabetes, type 2 diabetes, and gestational diabetes for women), cardiovascular disease (CVD) or cancer at and before the baseline for the dietary analyses.
* Participants who left more than 70 of the 131 food items blank on the baseline FFQ, reported unusual total energy intake levels (<3,347 or >17,573 kJ/day for men, and <2,092 or >14,644 kJ/day for women), or had missing baseline dietary information.
* Participants who only completed the baseline questionnaire.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Participant eligibility is based on self-representation of gender identity.
Study Population: The Nurses' Health Study (NHS) consisted of 121,700 female registered nurses enrolled in 1976. The NHSII was initiated in 1989 with the recruitment of 116,671 younger female registered nurses. The Health Professionals Follow-up Study (HPFS) was established in 1986 and was comprised of 51,529 US male health professionals.
Sampling Method: Non-Probability Sample
Enrollment: 289900 (Actual)
Dates: Start 1980-08 (Actual); Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Type 2 diabetes | Since 1976, with active follow-up
  Type 2 diabetes
Cardiovascular disease | Since 1976, with active follow-up
  Coronary heart disease and stroke
Mortality | Since 1976, with active follow-up
  Deaths due to various causes

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Belanger CF, Hennekens CH, Rosner B, Speizer FE. The nurses' health study. Am J Nurs. 1978 Jun;78(6):1039-40. No abstract available. PMID 248266
- [Result] Rimm EB, Giovannucci EL, Willett WC, Colditz GA, Ascherio A, Rosner B, Stampfer MJ. Prospective study of alcohol consumption and risk of coronary disease in men. Lancet. 1991 Aug 24;338(8765):464-8. doi: 10.1016/0140-6736(91)90542-w. PMID 1678444
- [Derived] Ma L, Liu G, Sampson L, Willett WC, Hu FB, Sun Q. Dietary glucosinolates and risk of type 2 diabetes in 3 prospective cohort studies. Am J Clin Nutr. 2018 Apr 1;107(4):617-625. doi: 10.1093/ajcn/nqy003. PMID 29635498
- See also: Nurses' Health Studies — http://www.nurseshealthstudy.org/